CLINICAL TRIAL: NCT01204632
Title: Cardiometabolic Risk, Obesity and Cardiovascular Disease in People With Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: MedStar National Rehabilitation Network (Other)
Responsible Party: Principal Investigator, Mark S. Nash, Ph.D., FACSM, Professor, University of Miami
Other Study IDs: TMP-MN-008
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to develop and field-test new tools for diagnosis and hazard assessment of cardiometabolic risk (CMR) in people with chronic spinal cord injury (SCI) and to advance the evidence base with much needed information on CMR and cardiovascular disease (CVD) burden in people with SCI. These data can be used to develop screening guidelines for early identification and prevention of CMR in SCI, as well as targeted approaches to primary disease management.

DETAILED DESCRIPTION:
Unlike current assessments utilizing lipid scores, the new system will be anchored in more reliable measurements of cardiovascular disease (CVD) burden using contemporary surrogate end points of coronary artery calcium (CAC) score, coronary CT angiography and carotid intima media thickness (CIMT). By the end of the 5-year funding cycle we will develop an updatable web-based cardiometabolic risk assessment tool (RISK) that will allow clinicians and SCI consumers to quantify risk for a cardiovascular sentinel event (stroke, non-fatal heart attack, or death) and will also provide a body mass index (BMI) table adjusted for SCI.

Specific Aims:

1. Examine the relationships among surrogates of cardiovascular disease burden in persons with SCI and established cardiometabolic risks.
2. Identify significant predictors of cardiometabolic risk (CMR) that are unique to persons with specific levels of SCI.
3. Develop and validate SCI CMR assessment tool (RISK) based on cardiometabolic risk scores.
4. Develop and validate an adjusted BMI table for SCI.

ELIGIBILITY:
Inclusion Criteria:

* traumatic spinal cord injury between C4 and T12
* have a motor complete injury as classified as American Spinal Injury Association Impairment Scale (AIS) grade A or B
* injury for more than 1 year
* no known history of traumatic brain injury, cardiovascular disease or diabetes
* not currently taking any medications to treat cardiovascular disease or diabetes
* have multiple (i.e., 2+) of the following cardiometabolic risk factors:

  1. fasting triglyceride > 150 mg/dL
  2. HDLC < 40 mg/dL
  3. hs-CRP > 3.0
  4. body fat (by DEXA) >25% for males and 33% for females

Exclusion Criteria:

* history of allergy or hypersensitivity to fish and/or nuts
* undergoing anticoagulant therapies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample of healthy persons with spinal cord injury
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2010-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Body composition | 1 visit
  The percent of muscle and fat in each participants' body will be measured by dual x-ray absorptiometry (DEXA) scan.

SECONDARY OUTCOMES:
Carotid Intima-Media Thickness | 1 visit
  Carotid intima-media thickness (IMT) measurements will be generated using B-mode external vascular ultrasound.
Coronary Artery Calcium | 1 visit
  Non-contrast cardiac CT will be used to measure coronary artery calcium, as the presence of any calcium detected in the coronary tree is diagnostic of atherosclerosis. The volume of calcium is quantified, providing a score of plaque burden analogous to a physiologic stress test. Coronary calcium scores directly correlate with risk of cardiac events, with higher scores indicating greater plaque burden and greater risk of cardiac events.
Atherosclerotic plaques | 1 visit
  Noninvasive CT angiography will be used in visualizing both calcified and non-calcified atherosclerotic plaques. This technique provides much finer anatomic detail and provides an opportunity to further identify latent atherosclerosis risk through the detection of both calcified and noncalcified atherosclerosis.
Area Under the Curve (AUC)for lipemia | 1 visit
  Lipemia is assessed by the AUC for triglycerides during an oral glucose tolerance test.
Area Under the Curve (AUC) for glycemia | 1 visit
  Glycemia is assessed by the AUC for glucose and insulin during an oral glucose tolerance test.
Area Under the Curve (AUC)for vascular inflammation | 1 visit
  The pro-atherogenic inflammatory mediators are AUCs for C-reactive protein and Interleukin-6 during an oral glucose tolerance test.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nash, PhD, Principal Investigator — University of Miami Miller School of Medicine, The Miami Project to Cure Paralysis
Locations (1):
- The Miami Project to Cure Paralysis, Miami, Florida, United States